CLINICAL TRIAL: NCT03709511
Title: A Randomized, Open-label, Controlled Trial on Perioperative Rehabilitation of Cardiac Valvular Surgery
Brief Title: Perioperative Rehabilitation of Cardiac Valvular Surgery
Acronym: PORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Chen, professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GDCR2017143H
Record Dates: First submitted 2018-02-26; First posted 2018-10-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Heart Valve Diseases; Pulmonary Complication
Keywords: Heart valve surgery; Rehabilitation; Physical exercise; Psycho-education
MeSH Terms: conditions — Heart Valve Diseases; Motor Activity | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Masking Description: Both the researchers and participants know which treatment is being administered(An open-label trial).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment Group (No Intervention): Participants in the control group will receive the usual care protocol. On the day of admission, a registered nurse in cardiac ward will provide operating skills of deep breathing, cough exercises, and incentive spirometry, then patients will be instructed to perform the respiratory exercise as much as they can during the hospitalization without supervision. These participants will not receive additional rehabilitation interventions, unless individual indications are present.
- Cardiac Rehabilitation Group (Active Comparator): The intervention group will receive the PORT protocol, contains education, IMT, ACBT, EM. Participants will be provided information about the cardiac surgery and adverse effect on postoperative recovery, and the importance of PORT program.
  An inspiratory threshold-loading device is used for IMT. Participants will be instructed to breathe in as forcefully as possible before slowly breathing out five times and then rest for one minute, followed by another set of five breaths. Patients will complete three sessions of ACBT consisting of breathing control, thoracic expansion exercises and forced expiratory techniques. The mobilization protocol will be performed via a progressive approach, consisting of 6 steps. EM will be personalized to each patient.
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — perioperative rehabilitation consists of education, inspiratory muscle training, active cycle of breathing techniques, and early mobilization.
  Arms: Cardiac Rehabilitation Group

SUMMARY:
Approximately 70,000 cardiac valve surgeries are performed in China every year. Although guidelines or consensus recommendations recommend perioperative rehabilitation after valve surgery, clinical studies are still lacking, especially for Chinese patients. The investigators hope to find out whether a comprehensive cardiac rehabilitation program can improve the postoperative mortality, complications and length of stay m as well as anxiety, depression and quality of life, after heart valve surgery. A singlecenter, randomized clinical trial, PORT study, aims to investigate whether cardiac rehabilitation in addition to usual care is superior to treatment as usual after heart valve surgery. The trial will randomly allocate 800 patients after inclusion screening, 1:1 intervention to control group, using central randomization, and blinded outcome assessment and statistical analyses. The intervention consists of rehabilitation education, inspiratory muscle training (IMT), active cycle of breathing techniques (ACBT), and early mobilization (EM). The primary outcome of this study will be a composite of in-hospital all-cause mortality, the incidence of postoperative pulmonary complications, and the ratio of postoperative hospitalization > 7 days. The secondary outcomes will be (1) SICU days of stay; (2) days of bed rest; (3) days of hospital length of stay; (4) all-cause death in 3 months; (5) anxiety measured by Generalized Anxiety Disorder scale (GAD-7) and depression measured by Patient Health Questionnaire-9 (PHQ-9) in 3 months. (6) quality of life measured by the Short Form 36 (SF-36) in 3 months.

DETAILED DESCRIPTION:
The PORT study is a randomized, open-label, controlled trial using assessor blinding and intention-to-treat analysis. To date, no high-quality study has prospectively examined the impact of perioperative CR in the Chinese population undergoing cardiac surgery. Thus, the PORT trial has been designed to address a cardiac rehabilitation study in line with the actual situation in China. The investigators have used the Standard Protocol Items: Recommendations for Intervention Trials (SPIRIT) guidelines in reporting this clinical trial.

Eligible patients are invited to a face-to-face meeting to confirm study eligibility and introduce the study objectives. The screened candidates will sign the written informed consent after they confirm their willingness to participate. Baseline data are collected subsequently. Then, the intervention group will receive perioperative rehabilitation interventions targeted at the optimization of the postoperative outcomes, This specialized approach, the PORT protocol, contains four key elements: education, inspiratory muscle training (IMT), active cycle of breathing techniques (ACBT), and early mobilization (EM). Patients will be evaluated during hospitalization for study outcomes and 3 months after surgery.

After collection of baseline data, central randomization is conducted on a web-based interface (http://crdms.echobelt.org/) using a computer-generated randomized treatment allocation schedule. The randomization is stratified based on patients' age (<60, 60-75, and >75 years), left ventricular ejection fraction (<40%, 40%-50%, and >50%), and lung function (GOLD stage 1, 2, 3 and 4) with a permuted scheme with blocks of varying sizes, which is concealed from the investigators to avoid selection bias. Thus, neither investigators and patients nor relatives can influence the group the patients are allocated. Personal information about potential and enrolled patients will be collected electronically and shared in a database accessible only within the project group for those responsible for patient inclusion, in order to protect confidentiality before, during, and after the trial.

The investigators are performing a randomized trial stating that the mean in the intervention and the control groups are the same with a power of 95%, and a type I error probability of 5%. Data from the pilot study (to be submitted) showed that the incidence in the primary endpoint was 13.56% (intervention group) versus 21.21% (control group). The inclusion of 400 participants is needed in the experimental intervention group, and 400 in the control group (a total of 800 participants) to be able to reject the null hypothesis. The trial will randomly allocate 800 patients, 1:1 intervention to the control group, using central randomization, blinded outcome assessment, and statistical analyses. The intervention consists of education, inspiratory muscle training (IMT), active cycle of breathing techniques (ACBT), and early mobilization (EM), intervention versus treatment as usual, with blinded outcome assessment.

ELIGIBILITY:
Inclusion criteria:

Aged from 18 to 75 years. Scheduled for elective mitral and/or aortic valve repair/replacement. New York Heart Association Classification (NYHA) I-III.

Exclusion criteria:

Complicated with preoperative endocarditis and/or pneumonia. Requiring emergency surgery. Enrolled in another clinical trial. Severe liver failure (Child-Turcotte-pugh classification ≥ B). Dialysis-dependent renal failure. Residual neurological and musculoskeletal impairment. Irregular vital signs (heart rate: < 40 or > 120 bpm at rest; blood pressure: systolic blood pressure > 200 mm Hg or diastolic pressure > 110 mm Hg; T: ≥ 38.5 or ≤ 36◦C; RR: >40 bpm; SpO2 ≤ 90%).

Unwilling or unable to sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
composite end point of in-hospital all-cause death, pulmonary complications and the ratio of postoperative hospitalization longer than 7 days. | Through hospitalization (up to 2 months)
  the composite of in-hospital all-cause death and pulmonary complications, such as pulmonary infection, postoperative hospitalization days.

SECONDARY OUTCOMES:
incidence of all-cause death in 3 months | 3 months
  incidence of all-cause death at 3-month follow-up.
Individualized Short Form-36 (SF-36) living quality Scores in 3 months | 3 months
  Scores from the self-administered SF-36 living quality questionnaire are measured. Higher mean scores reflect better outcomes.
length of ICU treatment | Through hospitalization (up to 2 months)
  total length of treatment at Intensive Care Unit
total length of in-hospital stays | Through hospitalization (up to 2 months)
  total length of in-hospital stays
length of bed rest | Through hospitalization (up to 2 months)
  length of bed rest Description: post-operative duration of bed rest until off-bed activity supervised by rehabilitation therapists.
Incidence of Treatment-Emergent Adverse Events [Emerging Arrhythmia or/and Muscle Injury or/and Acute Heart Failure] | Through hospitalization (up to 2 months)
  The evaluation of Treatment-Emergent Adverse Events during hospitalization: Emerging Arrhythmia or/and Muscle Injury or/and Acute Heart Failure.
Anxiety and depression in 3 months | 3 months
  anxiety measured by Generalized Anxiety Disorder scale (GAD-7) and depression measured by Patient Health Questionnaire-9 (PHQ-9) in 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou H, Liu F, Liu Y, He X, Ma H, Xu M, Wang H, Zhang G, Cai X, Chen JY, Guo L, Chen J. Protocol for the PORT study: short-term perioperative rehabilitation to improve outcomes in cardiac valvular surgery - a randomised control trial. BMJ Open. 2023 Dec 21;13(12):e074837. doi: 10.1136/bmjopen-2023-074837. PMID 38135333
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483